CLINICAL TRIAL: NCT01165398
Title: Comprehensive Evaluation of a Central Line Simulation Course
Status: Completed | Type: Observational
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Other Study IDs: 1-20090107
Record Dates: First submitted 2010-07-12; First posted 2010-07-19 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Infection
Keywords: Education; central lines; infections; complications; Bundles
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Residents, PAs, mid level providers: Lehigh Valley Health Network residents, physician assistants, and mid level providers who place central lines and attend the central lines simulation course

SUMMARY:
An estimated 250,000 cases of central line-associated bloodstream infections occur in US hospitals annually, and an estimated 30,000 to 62,000 patients die as a result, the marginal cost of which to the health-care system is approximately $25,000 per episode. Inconsistent and outdated clinical practices have been identified as key causative factors. In order to improve overall healthcare delivery and outcomes, current and future healthcare professionals need to complement their clinical skills with systems-based skills. Specific to the problems of central lines, during a 2005 chart review of institutional patient safety issues, a LVHN internal quality committee found multiple cases involving the insertion of central lines, including cases involving arterial placement and malposition. The internal quality committee review revealed that newer residents were primarily involved in these cases. As a result of the committee's findings and review of the literature, a standardized Central Line Access and Placement course was designed as part of the incoming residents'orientation process. This study's goal was to contribute to the knowledge-base of health professional education and to build a sustainable model for one set of learning and development interventions, with the expectation that findings will have broad relevance for patient safety initiatives, health professional training and development programs, and healthcare delivery improvement.

DETAILED DESCRIPTION:
Each year,"an estimated 250,000 cases of central line-associated bloodstream infections occur in U.S. hospitals, and an estimated 30,000 to 62,000 patients die as a result" (AHRQ 2008). The marginal cost to the health-care system is approximately $25,000 per episode (CDC 2002).Inconsistent and outdated clinical practices have been identified as key factors to this problem(5 Million Lives Campaign 2008). Subsequently, in order to improve overall healthcare delivery and outcomes, current and future healthcare professionals need to complement their clinical skills with systems-based skills such as: (a) delivering patient-centered care,(b) working in multidisciplinary care teams,(c) practicing evidence-based medicine,(d)focusing on quality improvement,and e)using information technology (IOM 2003).

Specific to the problems of central lines, during a February 2005 chart review of institutional patient safety issues, a LVHN internal quality committee found multiple cases involving the insertion of central lines, including cases involving arterial placement and malposition.The internal quality committee review revealed that newer residents were primarily involved in these cases. According to the literature, risk of central lines complication tends to decrease with operator experience (Runyon, 1986).A failed catheter placement attempt is one of the strongest predictors of subsequent complications (Haire & Lieberman, 1995). As a result of the committee's findings and review of the literature, a standardized Central Line Access and Placement course was designed as part of the incoming residents'orientation process.

Using Donald Kirkpatrick's Four-Level Evaluation model(Kirkpatrick and Kirkpatrick 2006) as a theoretical framework, this study analyzes the impact of a central lines simulation course on residents and mid-level providers' clinical performance and patient outcomes.It is the goal of this study to contribute to the knowledge-base of health professional education and to build a sustainable model for one set of learning and development interventions, with the expectation that findings will have broad relevance for patient safety initiatives, health professional training and development programs, and healthcare delivery improvement.

Care bundles are groupings of best practices with respect to a disease process that individually improve care, but when applied together result in substantially greater improvement.The science supporting each bundle component is sufficiently established to be considered the standard of care (5 Million Lives Campaign 2008).The central line bundle is a group of evidence-based interventions for patients with intravascular central catheters that, when implemented together, result in better outcomes than when implemented individually.The central line bundle has five key components:

1. Hand hygiene
2. Maximal barrier precautions
3. Chlorhexidine skin antisepsis
4. Optimal catheter site selection, with subclavian vein as the preferred site for non-tunneled catheters
5. Daily review of line necessity, with prompt removal of unnecessary lines Research Questions How does the quality of central line instruction relate to learner attitudes, knowledge, and compliance of the central line bundle? How do variations among course participants in the quality of central line instruction, knowledge of central lines, central line bundle compliance, and other factors relate to the complication and infection rates of their patients? How have central lines bundle compliance and central line-related complication and infection rates at LVHN changed over the past several years, and do those changes correspond to changes in policies and practice regarding central lines that have occurred since 2005? Objectives

1.Analyze the impact of a central line simulation course on learner, patient and business outcomes. 2.Incorporate 'standard of care' course improvements to enrich analysis of research. Hypotheses H0: There is no association among quality of central line instruction, learner knowledge, compliance of the central line bundle, complication and infection rates, and changes in policies and practice since 2005.

H1: There is an association among quality of central line instruction, learner knowledge, compliance of the central line bundle, complication and infection rates and changes in policies and practice since 2005.

Hc: There is a direct correlation among quality of central line instruction, learner knowledge, compliance of the central line bundle, and complication/infection rates.

Hk&b: There is a probably ratio among complication/infection rates from central lines based on variations in learner knowledge scores and bundle compliance.

Hp&p: There is a probability ratio among complication/infection rates from central lines based on changes in Lehigh Valley Health Network policies and practices over time (in months).

ELIGIBILITY:
Inclusion Criteria:

* Lehigh Valley Health Network residents, physician assistants, and nurse practitioners who place central lines and attend the central lines simulation course

Exclusion Criteria:

* Those residents, physician assistants, and nurse practitioners who place central lines and attend the central lines simulation course, but do not wish to participate in the audio taped focus groups

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lehigh Valley Health Network residents, physician assistants, and nurse practitioners who place central lines and attend the central lines simulation course
Sampling Method: Non-Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
How do variations among course participants in the quality of central line instruction, knowledge of central lines, central line bundle compliance, and other factors relate to the complication and infection rates of their patients? | At time of complication or infection
  To determine the extent to which ratings of faculty teaching performance, central lines knowledge test scores, performance check scores, and bundle compliance scores, along with variables from the operator database (e.g., Job, Program/Unit, Course Date, Approximate Number of Lines Placed, Number of and/or ICU rotations), relate to complication rates and infection rates.

SECONDARY OUTCOMES:
How does the quality of central line instruction relate to learner attitudes, knowledge, and compliance of the central line bundle? | At time of complication or infection
  To measure the relationship between course participants' rating of teaching performance against subscale and overall scores of the central lines knowledge test,and scores from the Performance Check Critical Action worksheet against the total compliance scores. Focus group data will be analyzed to identify perceptions, practices, power dynamics, and barriers to using the checklist and other patient safety protocols of the procedure.
How have central lines bundle compliance and central line-related complication/infection rates at LVHN changed, and do those changes correspond to changes in policies and practice regarding central lines? | At time of complication or infection
  Conduct a regression analysis utilizing time (in months) as the predicting variable and complication and infection rates as outcome variables.

CONTACTS AND LOCATIONS:
Overall Officials: Marna R. Greenberg, DO, Principal Investigator — Lehigh Valley Health Network
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AHRQ Awards $3 Million To Help Reduce Central Line-Associated Bloodstream Infections in Hospital ICUs. Press Release, October 1, 2008. Agency for Healthcare Research and Quality, Rockville, MD. http://www.ahrq.gov/news/press/pr2008/clabipr.htm
- [Background] O'Grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA. Guidelines for the prevention of intravascular catheter-related infections. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 Aug 9;51(RR-10):1-29. PMID 12233868
- [Background] Haire WD, Lieberman RP. Defining the risks of subclavian-vein catheterization. N Engl J Med. 1994 Dec 29;331(26):1769-70. doi: 10.1056/NEJM199412293312609. No abstract available. PMID 7605425
- [Background] Institute of Medicine, Health Profession Education Report. Washington, DC: National Academy Press, 2003.
- [Background] Kirkpatrick, D. Kirkpatrick, J. Evaluating Training Programs: The Four Levels. Third Edition, Berrett-Koehler Publishers, Inc. San Francisco, CA. 2006.
- [Background] Runyon BA. Paracentesis of ascitic fluid. A safe procedure. Arch Intern Med. 1986 Nov;146(11):2259-61. PMID 2946271
- [Background] 5 Million Lives Campaign. Getting Started Kit: Prevent Central Line Infections How-to Guide. Cambridge, MA: Institute for Healthcare Improvement; 2008. (Available at www.ihi.org)